CLINICAL TRIAL: NCT04981639
Title: Effects of Transabdominal Plane Block and Electrical Twitch Obtaining Intramuscular Stimulation on the Postoperative Pain in Cytoreductive Surgery and Hyperthermic Intra-peritoneal Chemotherapy (CRS and HIPEC): a Double-blind Randomized Control Trial
Brief Title: TAP and IMS for HIPEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3-2021-0032
Record Dates: First submitted 2021-07-25; First posted 2021-07-29 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Cytoreductive Surgery
Keywords: hyperthermic intra-peritoneal chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I (IVPCA) (Active Comparator): Intravenous patient controlled analgesia will be performed.
  Interventions: Procedure: IVPCA
- II (IVPCA+TAP) (Active Comparator): Intravenous patient controlled analgesia and transversus abdominis plane block will be performed.
  Interventions: Procedure: TAP
- III (IVPCA, IMS, and TAP) (Active Comparator): Intravenous patient controlled analgesia, transversus abdominis plane block, and intramuscular muscular stimulation will be performed.
  Interventions: Procedure: IMS

INTERVENTIONS:
Procedure: IVPCA — Intravenous patient controlled analgesia will be performed.
  Arms: I (IVPCA)
Procedure: TAP — Transversus abdominis plane block will be performed.
  Arms: II (IVPCA+TAP)
Procedure: IMS — Intramuscular electrical stimulation will be performed.
  Arms: III (IVPCA, IMS, and TAP)

SUMMARY:
It is important to decrease the postoperative pain in patients undergoing cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy. We will compare the Transversus abdominis plane block with the Transversus abdominis plane block plus intramuscular electrical stimulation in patients undergoing cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

-Patients who are able to do daily activity and walk independently.

Exclusion Criteria:

1. Patients with history of preoperative abdominal surgery
2. Patients who are unable to walk independently due to musculoskeletal disorder
3. Patients who are allergic to local anesthetics
4. Patients with chronic pain
5. Patients with pacemaker
6. Patients with endotracheal tube postoperatively
7. Patients with history of substance abuse
8. Pregnancy
9. Patients who are unable to communicate due to mental disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Pain score | At postoperative day 1
  Pain score will be measured using visual analogue scale (0: no pain, 10: worst imaginable pain) at postoperative day 1.

SECONDARY OUTCOMES:
Pain score | At postoperative day 2, 3, 5, 7, 14 and 28
  Pain score will be measured using visual analogue scale (0: no pain, 10: worst imaginable pain) at postoperative day 0, 2, 3, 5, 7, 14 and 28.
IVPCA consumption | At postoperative day 1, 2, and 3
  Intravenous patient controlled analgesia consumption will be measured at postoperative day 0, 1, 2, and 3.
Nausea will be evaluated using 2 point scale (yes, no) | At postoperative day 1, 2, 3, 5 and 7
  Nausea will be evaluated using 2 point scale (yes, no) at postoperative day 1, 2, 3, 5 and 7.
Vomiting will be evaluated using 2 point scale (yes, no) | at postoperative day 1, 2, 3, 5 and 7.
Peak cough flow | At postoperative day -1, 4, 7, 14, and 28
  Peak cough flow will be evaluated at postoperative day -1, 4, 7, 14, and 28.
Gait speed | day -1, 4, 7, 14, and 28
  Gait speed will be evaluated at postoperative day -1, 4, 7, 14, and 28.
Quality of life will be evaluated using QoR40 questionnaire (0-200) | At postoperative day 4 and 7
  Quality of life will be evaluated using QoR40 questionnaire (0-200) at postoperative day 4 and 7.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeveranceHospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HC, Park J, Oh J, Kim M, Park EJ, Baik SH, Song Y. Analgesic effects of combined transversus abdominis plane block and intramuscular electrical stimulation in patients undergoing cytoreductive surgery followed by hyperthermic intraperitoneal chemotherapy: a randomized controlled trial. Int J Surg. 2023 May 1;109(5):1199-1207. doi: 10.1097/JS9.0000000000000383. PMID 36999805